CLINICAL TRIAL: NCT02598778
Title: Comparing Chlorhexidine Gluconate Rinse, Sodium Fluoride Rinse, Water Rinse, and Chewing Gum in Regard to Streptococcus Mutans Reduction
Brief Title: Comparing Mouth Rinses (and Chewing Gum) in Regard to Streptococcus Mutans Reduction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued early due to time constraints and lack of selectivity in agar used in the identification of the target (Streptococcus mutans). Only 12 participants out of a planned 40 were enrolled.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Nuntiya Kakanantadilok, Asst. Prof. Dentistry, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-5583
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Dental Caries
Keywords: Streptococcus Mutans; Saliva
MeSH Terms: conditions — Dental Caries | interventions — chlorhexidine gluconate; Sodium Fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Chlorhexidine gluconate (0.12%) (Active Comparator): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Interventions: Drug: Chlorhexidine gluconate (0.12%)
- Sodium Fluoride (0.05%) (Active Comparator): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Interventions: Drug: Sodium Fluoride (0.05%)
- Paraffin wax chewing gum (sugar-free) (Placebo Comparator): A food product. Minimum of 2 minutes of chew time prior to salivary sample being obtained.
  Interventions: Other: Paraffin wax chewing gum (sugar-free)
- Deionized water (Placebo Comparator): Water that has had the majority of its ions removed.
  Interventions: Other: Deionized water

INTERVENTIONS:
Drug: Chlorhexidine gluconate (0.12%) — 30 second oral rinse of 10mL of solution
  Other Names: Peridex
  Arms: Chlorhexidine gluconate (0.12%)
Drug: Sodium Fluoride (0.05%) — 30 second oral rinse of 10mL of solution
  Other Names: ACT brand anticavity mouthrinse
  Arms: Sodium Fluoride (0.05%)
Other: Paraffin wax chewing gum (sugar-free) — Approximately two minutes of chew time
  Arms: Paraffin wax chewing gum (sugar-free)
Other: Deionized water — 30 second oral rinse of 10mL of solution
  Arms: Deionized water

SUMMARY:
This study compared four mouth rinses/chews for their ability to reduce Streptococcus Mutans after usage. The four that were compared were chlorhexidine gluconate (0.12%), sodium fluoride (0.05%), paraffin wax chewing gum (sugar free), and deionized water. The paraffin wax chewing gum replaced the originally planned coconut oil and served as a placebo comparator.

DETAILED DESCRIPTION:
The study was a randomized controlled clinical trial, unblinded. After obtaining consent and assent, respectively, and following review of medical history with regard to inclusion/exclusion criteria, if the participant met eligibility criteria, the participant was randomly assigned to one of four groups being studied: chlorhexidine gluconate (0.12%), sodium fluoride (0.05%), paraffin wax chewing gum (sugar-free) or deionized water with a randomization ratio of 1:1:1:1. A pre rinse/chew salivary sample was obtained by having the participant spit into a sterile test tube. The participant then either rinsed with 10mL of the assigned rinse for a timed 30 seconds and expectorated, or chewed paraffin wax chewing gum for 2 minutes. A post rinse/chew salivary sample was taken similarly to the pre rinse/chew sample. The samples were transported to a microbiology lab for incubation and quantitative analysis of Streptococcus Mutans. Morphological identification of the bacterial colonies was then confirmed using Matrix Assisted Laser Desorption/Ionization Time of Flight (MALDI-TOF) mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the dental clinic for routine dental treatment (including recall exams, new patient exams, and operative appointments) who are American Society of Anesthesia (ASA) class I or II
* Cooperative patients classified as 3 or 4 according to the Frankl Behavioral Rating Scale,
* No known allergies or sensitivities to products or ingredients being tested
* Had untreated cavities
* Nothing to eat/drink for 1 hour prior to dental appointment

Exclusion Criteria:

* Patients who are ASA class III, IV, V or VI
* Known allergies or sensitivities to any of the mouth rinses or any of the ingredients in the mouth rinses to be tested
* Non-English speaking parent/participant
* Patient presenting to the clinic as a walk in or emergency appointment
* Patient experiencing any pain or sensitivity
* Precooperative or uncooperative behavior or behavior classified as 1 or 2 according to the Frankl Behavioral Rating Scale

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nuntiya Kakanantadilok, DMD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine Gluconate (0.12%): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Chlorhexidine gluconate (0.12%): 30 second oral rinse expectorate of 10mL of solution
- Sodium Fluoride (0.05%): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Sodium Fluoride oral rinse (0.05%): 30 second oral rinse expectorate of 10mL of solution
- Paraffin Wax Chewing Gum (Sugar-free): A food product serving as placebo.
  Paraffin wax chewing gum (sugar-free): 2 minutes of chew time prior to salivary sample being obtained
- Deionized Water: Water that has had the majority of its ions removed.
  Deionized water: 30 second oral rinse expectorate of 10mL of solution
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate (0.12%) | Sodium Fluoride (0.05%) | Paraffin Wax Chewing Gum (Sugar-free) | Deionized Water
Started | 2 | 4 | 4 | 2
Completed | 2 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sodium Fluoride (0.05%): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Sodium Fluoride (0.05%): 30 second oral rinse expectorate of 10mL of solution
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Gluconate (0.12%) | Sodium Fluoride (0.05%) | Paraffin Wax Chewing Gum (Sugar-free) | Deionized Water | Total
Number analyzed (Participants) | 2 | 4 | 4 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 4 | 2 | 12
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were not collected for Sex/Gender
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 4 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Salivary Streptococcus Mutans Levels After 30 Second Oral Rinse Time (Chlorhexidine Gluconate, Sodium Fluoride, or Deionized Water) or 2 Minute Chew Time (Paraffin Wax Chewing Gum)
Description: Oral salivary sample obtained and plated on MSB (mitis salivarius-bacitracin) agar petri dish to determine Streptococcus mutans (S. mutans) levels.
  Values in each row in the Outcome Measure Data Table represent percentage change (increase denoted by positive number, decrease denoted by negative number) in S. mutans colonies from baseline (pre rinse/chew) sample for a single participant within that particular Arm/Group. Row titles have been arbitrarily identified as 'First Participant', 'Second Participant', 'Third Participant' and 'Fourth Participant.' No values are shown for 'Third Participant' and 'Fourth Participant' for the Chlorhexidine gluconate (0.12%) and Deionized water Arm/Group since only 2 participants were enrolled within each group. One result is obtained from each pre and post sample combination (percentage change).
Time Frame: Sample obtained at baseline (pre rinse/chew) and immediately after treatment (post rinse/chew). Timed for 30 seconds (oral rinses) or 2 minutes (chewing gum)
Population: 1 pre (baseline) and post sample was collected and analyzed from each participant. As such, there were 2 pre and 2 post samples for the Chlorhexidine gluconate Arm/Group, 4 pre and 4 post samples for the Sodium Fluoride Arm/Group, 4 pre and 4 post samples for the Paraffin wax chewing gum Arm/Group, and 2 pre and 2 post samples for the Deionized water Arm/Group. Values in Outcome Measure Data table reflects percentage change (increase/decrease) in S. mutans colonies from pre (baseline) to post.
Measure: Number; unit: Percentage change in S. mutans colonies
Units Other Than Participants: Samples
Arm/Group | Chlorhexidine Gluconate (0.12%) | Sodium Fluoride (0.05%) | Paraffin Wax Chewing Gum (Sugar-free) | Deionized Water
Number analyzed (Participants) | 2 | 4 | 4 | 2
Number analyzed (Samples) | 2 | 4 | 4 | 2
Percentage change in S. mutans colonies
  First Participant: number analyzed (Participants) | 1 | 1 | 1 | 1
  First Participant: number analyzed (Samples) | 1 | 1 | 1 | 1
  First Participant | -100 | -75 | 53.13 | -39.29
  Second Participant: number analyzed (Participants) | 1 | 1 | 1 | 1
  Second Participant: number analyzed (Samples) | 1 | 1 | 1 | 1
  Second Participant | -100 | -100 | 88.89 | -46.15
  Third Participant: number analyzed (Participants) | 0 | 1 | 1 | 0
  Third Participant: number analyzed (Samples) | 0 | 1 | 1 | 0
  Third Participant |  | -100 | 161.54 |
  Fourth Participant: number analyzed (Participants) | 0 | 1 | 1 | 0
  Fourth Participant: number analyzed (Samples) | 0 | 1 | 1 | 0
  Fourth Participant |  | -100 | 176.26 |

ADVERSE EVENTS:
Time Frame: From the initiation of oral rinse/chew to the time of expectoration/spit (30 seconds - 2 minutes)
Groups:
- Chlorhexidine Gluconate (0.12%): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Chlorhexidine gluconate (.12%): 30 second oral rinse expectorate of 10mL of solution
- Sodium Fluoride (0.05%): An oral rinse given to pediatric patients in routine practice within the standard of care.
  Sodium Fluoride (.05%): 30 second oral rinse expectorate of 10mL of solution
Arm/Group | Chlorhexidine Gluconate (0.12%) | Sodium Fluoride (0.05%) | Paraffin Wax Chewing Gum (Sugar-free) | Deionized Water
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes